CLINICAL TRIAL: NCT03316131
Title: Quantifying Uric Acid Excretion With RDEA3170, Febuxostat and Dapagliflozin
Brief Title: A Study to Assess the Effect of Intensive Uric Acid (UA) Lowering Therapy With RDEA3170, Febuxostat, Dapagliflozin on Urinary Excretion of UA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Contract Research Organization: USA (Unknown); PAREXEL Early Phase Clinical Unit Baltimore (Unknown); PAREXEL Early Phase Clinical Unit-Los Angeles (Unknown); Clinical Laboratory: USA (Unknown); Harbor Hospital Laboratory (Unknown); GenX Laboratories Inc. (Unknown); Analytical Laboratory (Pharmacokinetic Sample Analysis): USA (Unknown); Covance Bioanalytical Services, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5495C00001
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2019-07-18 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Asymptomatic Hyperuricemia
Keywords: Gout; Uric acid; Hyperuricemia; Asymptomatic gout; Febuxostat; Dapagliflozin; Uric acid transporter 1 (URAT1) Inhibitor; Xanthine Oxidase Inhibitor; Sodium-glucose cotransporter 2 (SGLT2) Inhibitor
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — verinurad; Febuxostat; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The pharmacokineticist will remain blinded during the study conduct, unless otherwise required based on study findings. The pharmacokineticist will be unblinded to perform the final PK analyses after all patients have completed the study, final bioanalytical results are available and all required study data are considered clean. This may occur before database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Randomized patients will receive orally once daily fixed dose of the following drugs:
  verinurad + febuxostat + dapagliflozin;
  Interventions: Drug: Verinurad; Drug: Febuxostat; Drug: Dapagliflozin
- Treatment B (Experimental): Randomized patients will receive orally once daily fixed dose of the following drugs:
  verinurad + febuxostat + dapagliflozin matched placebo
  Interventions: Drug: Verinurad; Drug: Febuxostat; Other: Dapagliflozin matched placebo

INTERVENTIONS:
Drug: Verinurad — Randomized patients will receive orally once daily fixed dose of verinurad in 2 treatment sequences AB or BA for 7 consecutive days. Treatment A: verinurad + febuxostat + dapagliflozin; Treatment B: verinurad + febuxostat + placebo
  Other Names: RDEA3170
Drug: Febuxostat — Randomized patients will receive orally once daily fixed dose of febuxostat in 2 treatment sequences AB or BA for 7 consecutive days. Treatment A: verinurad + febuxostat + dapagliflozin; Treatment B: verinurad + febuxostat + placebo
  Other Names: ULORIC
Drug: Dapagliflozin — Randomized patients will receive orally once daily fixed dose of dapagliflozin in 2 treatment sequences AB or BA for 7 consecutive days. Treatment A: verinurad + febuxostat + dapagliflozin; Treatment B: verinurad + febuxostat + placebo
  Other Names: FARXIGA
  Arms: Treatment A
Other: Dapagliflozin matched placebo — Randomized patients will receive orally once daily fixed dose of dapagliflozin matched placebo in 2 treatment sequences AB or BA for 7 consecutive days. Treatment A: verinurad + febuxostat + dapagliflozin; Treatment B: verinurad + febuxostat + placebo
  Arms: Treatment B

SUMMARY:
This is a randomized, placebo controlled, double-blind, 2-way crossover study conducted on asymptomatic hyperuricemic patients. The core study consists of screening period, 2 treatment periods (verinurad + febuxostat + dapagliflozin/placebo) and follow-up visit

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, double-blind, 2-way crossover study to assess the effect of intensive UA lowering therapy with verinurad (RDEA3170), febuxostat, and dapagliflozin on urinary excretion of UA, in asymptomatic hyperuricemic patients. Thirty-six asymptomatic hyperuricemic patients aged 18 to 65 years (inclusive) will be enrolled into this study at 2 study centers. Twenty-four patients have been enrolled and completed the study to date. Due to inadequate urine sampling, 12 additional patients were included to ensure an adequate sample size (at least 20 evaluable patients) to evaluate the effects of intensive UA lowering with verinurad, febuxostat and dapagliflozin on urinary excretion of UA. With 24 completers available during the interim analysis, this will provide for a total sample size of 36 evaluable patients.

Before any study specific assessments are performed, potential patients must provide informed consent. Each patient will undergo the below mentioned visits:

* A Screening period of maximum 28 days;
* Two treatment periods during which patients will be resident in the Clinical Unit from Day -2 to Day 1 and from Day 6 to Day 8; and
* A Follow-up Visit within 14 to 28 days after the first administration of Investigational Medicinal Product (IMP) in Treatment Period 2.

On Day -2 of Treatment period 1, patient will be randomized (1:1) to 1 of 2 treatment sequences (AB or BA). Each randomized patient will receive orally once daily fixed dose of the below mentioned 2 treatments for 7 consecutive days (1 treatment per treatment period).

* Treatment A: Verinurad + febuxostat + dapagliflozin
* Treatment B: Verinurad + febuxostat + placebo For each treatment period, baseline measurements will be performed. On Day 1, after all dosing and all assessments have been performed, patients will receive instruction to administer the IMP at home once daily in the morning from Day 2 to Day 6 and the IMP will be dispensed for home dosing. Patients will return to the Clinical Unit on Day 6 and will be residential in the Clinical Unit from Day 6 to Day 8.

Treatment Period 1 and Treatment Period 2 will be separated by a washout period of 7 to 21 days.

Patients will return to the Clinical Unit for a Follow-up Visit, 14 to 28 days after Day 1 of Treatment Period 2.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old
2. Asymptomatic hyperuricemia (sUA > 6.0 mg/dL)
3. Body mass index between 18 and 35 kg/m2 inclusive and weight at least 50 kg and no more than 150 kg
4. Females must be non-pregnant, as well as post-menopausal or willing to use an acceptable method of contraception during the study.

Exclusion Criteria:

1. History of any clinically significant disease or disorder putting the patient at risk during the study, or influencing study results or ability to participate in the study
2. eGFR* < 45 mL/minute/1.73 m2 at Screening.
3. Type 2 diabetes mellitus with HbA1c >8%.
4. History of diabetic ketoacidosis, hyperosmolar non-ketotic coma, gout, or alcohol or drug abuse.
5. Ongoing treatment with an SGLT2-inhibitor, a URAT1-inhibitor, and/or a xanthine oxidase inhibitor.
6. Positive test for hepatitis B, hepatitis C or HIV.
7. Use of any medications in the 2 weeks preceding first administration of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stack AG, Han D, Goldwater R, Johansson S, Dronamraju N, Oscarsson J, Johnsson E, Parkinson J, Erlandsson F. Dapagliflozin Added to Verinurad Plus Febuxostat Further Reduces Serum Uric Acid in Hyperuricemia: The QUARTZ Study. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2347-e2356. doi: 10.1210/clinem/dgaa748. PMID 33075806
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14659&filename=AstraZeneca%20D5495C00001%20study%20(PXL236229)_SAP%20Amendment_1.0_16July2018_Redacted.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14659&filename=D5495C00001-CSP_amendment-3-signed_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at two study centres: Baltimore and Los Angeles. The date of the first subject visit was 25 Oct 2017 and the date of the last subject last visit was 19 Jul 2018. A total of 36 adults asymptomatic hyperuricemic patients were included into this study.
Pre-assignment Details: Patients who provided informed consent underwent screening procedures within the 28 days. Patients returned to the Clinical Unit on Day -2 of Treatment Period 1 and were randomized (1:1) to two treatment sequences ( treatment AB or BA).
Groups:
- Treatment Sequence A+B: Each patient received orally once daily dose of 9 mg verinurad + 80 mg febuxostat + 10 mg dapagliflozin (Treatment A). Each patient randomized to treatment A in period 1 received Treatment B in period 2 as this is 2-way crossover study
- Treatment Sequence B+A: Each patient received orally once daily dose of 9 mg verinurad + 80 mg febuxostat + placebo (Treatment B). Each patient randomized to treatment B in period 1 received Treatment A in period 2 as this is 2-way crossover study
Period: Treatment Period 1
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Protocol deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Each patient received orally once daily dose of 9 mg verinurad + 80 mg febuxostat + 10 mg dapagliflozin/placebo. Each patient randomized to treatment A in period 1 received Treatment B in period 2 and each patient randomized to treatment B in period 1 received Treatment A in period 2
Arm/Group | All Subjects
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 14
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Urinary Excretion of Uric Acid (UA) on Day 7
Description: Change from baseline in peak UA excretion during the first 8 hours on Day 7 of treatment to assess the effects of intensive UA lowering therapy with verinurad, febuxostat and dapagliflozin. Urine sample was collected in hourly intervals, and the highest amount of UA excreted in any interval was designated as peak UA excretion for each patient and treatment period.
Time Frame: On Day -1 and Day 7 of each treatment period
Population: Protocol Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams (mg)
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
milligrams (mg) | -12.87 [-21.03 to -4.70] | -13.15 [-21.31 to -4.98]
Statistical Analysis 1: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Test type: Other; Mean Difference (Net) = 0.28, 95% CI 2-sided [-8.67 to 9.22]

2. Primary Outcome: Change From Baseline in Plasma Concentration (Cmax) on Day 7
Description: Cmax assessment for Verinurad, M1, and M8 following daily oral administration of verinurad and febuxostat with and without dapagliflozin
Time Frame: On Treatment Period 1 and 2: Day 7 (Pre-dose and 15 minutes, 30 minutes, 1 hour, 1.5, 2, 3, 4, 8, 12 and 24 hours post-dose)
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
ng/mL
  Verinurad: number analyzed (Participants) | 35 | 36
  Verinurad | 17.52 (45.87) | 15.26 (52.48)
  M1: number analyzed (Participants) | 35 | 36
  M1 | 25.28 (41.55) | 25.61 (57.24)
  M8: number analyzed (Participants) | 35 | 36
  M8 | 18.45 (35.45) | 18.42 (44.36)
Statistical Analysis 1: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for Verinurad; Test type: Other; Geometric mean ratio = 1.14, 90% CI 2-sided [1.03 to 1.25]
Statistical Analysis 2: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for M1; Test type: Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.88 to 1.07]
Statistical Analysis 3: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for M8; Test type: Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.91 to 1.08]

3. Primary Outcome: Change From Baseline in Area Under Plasma Concentration Time Curve From Time Zero to the Time of Last Measurable Concentration (AUClast) on Day 7
Description: AUClast assessment for Verinurad, M1, and M8 following daily oral administration of verinurad and febuxostat with and without dapagliflozin
Time Frame: as for outcome 2
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h∙ng/mL
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
h∙ng/mL
  Verinurad: number analyzed (Participants) | 35 | 36
  Verinurad | 149.1 (37.79) | 141.0 (44.90)
  M1: number analyzed (Participants) | 35 | 36
  M1 | 212.7 (42.74) | 221.3 (49.13)
  M8: number analyzed (Participants) | 35 | 36
  M8 | 174.2 (34.57) | 176.5 (36.85)
Statistical Analysis 1: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for Verinurad; Test type: Other; Geometric mean ratio = 1.06, 90% CI 2-sided [1.00 to 1.13]
Statistical Analysis 2: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for M1; Test type: Other; Geometric mean ratio = 0.96, 90% CI 2-sided [0.90 to 1.02]
Statistical Analysis 3: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for M8; Test type: Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.94 to 1.04]

4. Secondary Outcome: Change From Baseline in Urinary Excretion of Serum UA (sUA) on Day 7
Description: Change from baseline in sUA to assess the intensive UA lowering effect of RDEA3170, febuxostat and dapagliflozin by evaluating the sUA levels after 7 days of treatment.
Time Frame: At Day -1 and Day 7
Population: Pharmacodynamic Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
umol/L | -327.161 [-352.559 to -301.762] | -264.851 [-290.060 to -239.643]

5. Secondary Outcome: Change From Baseline in Time to Reach Maximum Observed Concentration (Tmax) on Day 7
Description: tmax assessment for Verinurad, M1, and M8 following daily oral administration of verinurad and febuxostat with and without dapagliflozin
Time Frame: as for outcome 2
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
hour
  Verinurad: number analyzed (Participants) | 35 | 36
  Verinurad | 4.00 [2.00 to 8.00] | 4.00 [3.00 to 8.08]
  M1: number analyzed (Participants) | 35 | 36
  M1 | 4.00 [2.00 to 8.00] | 4.00 [3.00 to 4.03]
  M8: number analyzed (Participants) | 35 | 36
  M8 | 4.00 [3.00 to 8.02] | 4.00 [3.00 to 8.08]

6. Secondary Outcome: Change From Baseline in Time of Last Measurable Concentration (Tlast) on Day 7
Description: tlast assessment for Verinurad, M1, and M8 following daily oral administration of verinurad and febuxostat with and without dapagliflozin
Time Frame: as for outcome 2
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
hour
  Verinurad: number analyzed (Participants) | 35 | 36
  Verinurad | 24.00 [23.85 to 24.47] | 24.00 [23.22 to 24.40]
  M1: number analyzed (Participants) | 35 | 36
  M1 | 24.00 [23.85 to 24.47] | 24.00 [23.22 to 24.40]
  M8: number analyzed (Participants) | 35 | 36
  M8 | 24.00 [23.85 to 24.47] | 24.00 [23.22 to 24.40]

7. Primary Outcome: Change From Baseline in Area Under Plasma Concentration Time Curve Over a Dosing Interval (24 Hours) (AUCτ) on Day 7
Description: AUCτ assessment for Verinurad, M1, and M8 following daily oral administration of verinurad and febuxostat with and without dapagliflozin
Time Frame: as for outcome 2
Population: Pharmacokinetic Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h∙ng/mL
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
Number analyzed (Participants) | 36 | 36
h∙ng/mL
  Verinurad: number analyzed (Participants) | 35 | 36
  Verinurad | 149.0 (37.84) | 140.9 (44.90)
  M1: number analyzed (Participants) | 35 | 36
  M1 | 212.6 (42.78) | 221.1 (49.13)
  M8: number analyzed (Participants) | 35 | 36
  M8 | 174.1 (34.59) | 176.3 (36.81)
Statistical Analysis 1: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for Verinurad; Test type: Other; Geometric mean ratio = 1.06, 90% CI 2-sided [1.00 to 1.13]
Statistical Analysis 2: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for M1; Test type: Other; Geometric mean ratio = 0.96, 90% CI [0.90 to 1.02]
Statistical Analysis 3: Comparison: Treatment Sequence A+B vs Treatment Sequence B+A; Treatment A/Treatment B, for M8; Test type: Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.94 to 1.04]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of randomization throughout the treatment period up to and including the Follow-up Visit. Serious adverse events were recorded from the time of informed consent.
Description: From screening (Day -28) to follow-up (Day 23)
Arm/Group | Treatment Sequence A+B | Treatment Sequence B+A
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 7/35 | 5/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Sequence A+B (N=35) | Treatment Sequence B+A (N=36)
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Catheter Site Pain (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Vessel Puncture Site Haematoma (General disorders) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Eyelid Injury (Injury, poisoning and procedural complications) | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The initial plan was to recruit 24 patients, but due to difficulties in determining the peak urinary uric acid excretion in 11 patients, it was decided to include 12 additional patients to ensure adequate sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03316131/SAP_000.pdf
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT03316131/Prot_001.pdf